CLINICAL TRIAL: NCT06733636
Title: SPLENDOR-OA; Scents of Progress: Leveraging a Novel Device for Olfactory Training in Older Adults
Brief Title: Scents of Progress: Leveraging a Novel Device for Olfactory Training in Older Adults
Acronym: SPLENDOR-OA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00467494
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Olfactory Dysfunction; Smell Loss; Anosmia; Hyposmia
Keywords: Olfactory Dysfunction; Olfactory Training; Smell Training; Smell Training Device; Smell Loss; Anosmia; Hyposmia
MeSH Terms: conditions — Anosmia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Olfactory Training (Experimental): Participants will receive the ScentCare olfactory training device, which includes eight encapsulated scents: Eucalyptus, Cinnamon, Lemon, Coffee, Campfire, Cherry, Vanilla, and Lavender. To guide the participant in using the device, participants will have access to either a web-based application or a booklet, depending on the participant's preference. These resources will provide instructions on how to perform the smell training effectively. The training will be conducted twice daily over a period of three months.
  Interventions: Other: ScentCare (Olfactory Training Device)
- Control Arm (Sudoku Puzzles) (Other): Participants will be asked to complete sudoku puzzles twice daily over a period of three months.
  Interventions: Other: Sudoku Puzzles

INTERVENTIONS:
Other: Sudoku Puzzles — Sudoku puzzles of consistent and regular difficulty
  Arms: Control Arm (Sudoku Puzzles)
Other: ScentCare (Olfactory Training Device) — ScentCare is a smell training device with eight encapsulated scents housed in separate compartments and is contained using a charcoal filter, which will be dispersed in the base of our device to prevent smell contamination in the user's environment. The outer casing contains an opening that can be manually rotated to line up with the casing on each scent. This is facilitated by a rod in the center of the device, which serves as the axis of rotation. By pressing the capsule, the desired scent is released through a hole in the casing, similar to the mechanism of a pen. The user presses the compartment back downwards into the casing when done. The ScentCare mobile application offers clear instructions for at-home smell training and testing, with features like scent randomization to prevent users from getting accustomed to a specific order. It provides detailed guidance on device use and allows users to schedule sessions and receive daily reminders, ensuring a structured training regimen.
  Arms: Olfactory Training

SUMMARY:
The goal of this clinical trial is to learn if ScentCare, a novel olfactory training device and accompanying companion web-based application, will lead to improved olfactory and well-being outcomes in elderly patients with Olfactory Dysfunction (OD). The main question it aims to answer is:

- What effect does the olfactory training device (ScentCare) and accompanying companion web-based application have on olfaction?

Researchers will compare ScentCare to solving Sudoku puzzles to see the effects of olfactory training using this novel device on olfaction. Previous studies have used Sudoku puzzles when studying the effect of smell training. Since smell training is thought to work by stimulating and engaging higher order cognition, Sudoku is a suitable activity for participants in the control group since it serves as a correlate with similar degree of stimulation.

Participants will:

* Use ScentCare (intervention) or solve Sudoku puzzles (control) twice daily for 3 months.
* Visit the clinic twice, once upon enrollment and once three months later.
* Complete a formal smell test using Sniffin' Sticks smell test at the beginning of the study and again at the end of the study (3 months) during the initial and follow up visit.
* Complete questionnaires at the beginning of the study and again at the end of the study (3 months) during the initial and follow up visit.

DETAILED DESCRIPTION:
This research is being done to better understand the efficacy of an investigational device and its companion phone application (together called "ScentCare") in treating olfactory dysfunction.

Although the sense of smell is commonly overlooked, it is a unique and special human sensory function that has implications for quality of life, such as the enjoyment of food and nutrition or the ability to perceive dangers, such as smoke or noxious fumes. Although smell training is a well-established rehabilitation treatment for people with olfactory dysfunction (OD) or loss of smell, no standardized smell training method is currently available. Thus, the investigators invented a device and companion phone app that standardizes and compiles smell training. The investigators are seeking data on how to improve the device and its efficacy in general.

This study will have participants complete formal smell testing prior to using the ScentCare or Sudoku daily for three months and after the completion of the intervention. Participants will also answer a survey (questionnaires asked will include olfactory specific qualify of life assessment, cognitive assessment, depression assessment, anxiety assessment, device use and compliance) upon enrollment and after completion of the intervention (3 months follow up).

Once enrolled, participants will be randomized to either the "experimental" or "control" group. Participants in the experimental group will be given an olfactory training device and instructions for the smartphone-based olfactory training application. This olfactory training device consists of a hand-held rotating wheel with 8 individual scent chambers allowing personalized exposure to odorants (smells) according to the training app's instructions. If the participant does not have a smartphone, the participant will be given a training booklet with corresponding cues and instructions. Twice daily, 5-minute training sessions will be completed for 3 months. Participants in the control group will not undergo olfactory training but will be asked to complete sudoku puzzles for the same duration as the training for the experimental group.

After three months of either smell training with ScentCare or completing Sudoku puzzles, participants will be re-evaluated using the Sniffin' Sticks test and the same surveys to assess the impact of the intervention. Results will be compared between the two groups. Additionally, participants in the ScentCare group will provide feedback on the device's feasibility, ease of use, and overall effectiveness to inform its potential for broader application.

ELIGIBILITY:
Inclusion Criteria:

* Adults 60 years of age or older.
* English-speaking patients.
* Patients with a diminished or lost sense of smell.
* Patients who have not done smell training before

Exclusion Criteria:

* Patients who are sensitive to any of the scents used in the study.
* Patients with a diagnosis of congenital anosmia.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in olfaction as assessed by Sniffin' Sticks olfactory testing kit | Baseline and 3 months
  Changes in olfaction between the two groups will be assessed using Sniffin' Sticks olfactory testing. The main outcome is a cumulative Threshold, Discrimination, and Identification (TDI) score, where a TDI score above 30.5 is considered normal, between 30.5 and 16 indicates hyposmia (reduced smell), and below 16 signifies anosmia (complete loss of smell).

SECONDARY OUTCOMES:
Change in peripheral olfaction as assessed by Sniffin' Sticks olfactory testing kit | Baseline and 3 months
  Changes in peripheral olfaction between the two groups will be assessed using Sniffin' Sticks. Sniffin's Sticks tests olfactory function in three domains: threshold, discrimination, and identification. Threshold testing allows for peripheral olfaction testing. The most dilute concentration of odorant that the participant is able to reliably detect is determined. Score ranges between 1 and 16, with higher score indicating better peripheral olfaction.
Change in central olfaction as assessed by Sniffin' Sticks olfactory testing kit | Baseline and 3 months
  Changes in central olfaction between the two groups will be assessed using Sniffin' Sticks. Sniffin's Sticks tests olfactory function in three domains: threshold, discrimination, and identification. The discrimination and identification tests allow for central olfaction testing. In discrimination testing, the participant is evaluated on their ability to discern the unique scent among three scented sticks. In identification testing, the patient names the smell using a multiple choice form which offers four options for every scented stick, only one of which is correct.
  Both tests have scores ranging between 0 and 16, with higher scores indicating better central olfaction.
Change in olfactory specific Quality of Life as Assessed by the Questionnaire of Olfactory Disorders-Negative Statements (QOD-NS) | Baseline and 3 months
  Changes in overall olfactory wellbeing between the two groups will be assessed using Quality of life (QoL) assessment (Questionnaire of Olfactory Disorders-Negative Statements (QOD-NS). This instrument consists of 17 negative statements graded from 0 to 3 for a maximum score range of 0-51 (higher scores reflect worse QOL). The QOD-NS has 4 distinct factor domains, broadly categorized as those that relate to eating, anxiety, social interactions, and annoyance.
Change in overall cognition as assessed by the Montreal Cognitive Assessment (MoCA) test | Baseline and 3 months
  Changes in overall cognition will be assessed between the two groups using Montreal Cognitive Assessment (MoCA) test which is a rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. This test involves memorizing a short list of words, naming objects shown in pictures, copying shapes and performing other tasks. The test is scored out of a maximum of 30 points, and the results are interpreted as follows:
  26 or higher: Normal cognitive health; 18-25: Mild cognitive impairment (MCI); 10-17: Moderate cognitive impairment; Less than 10: Severe cognitive impairment
Change in overall anxiety as assessed by the General Anxiety Disorder Questionnaire-7 (GAD-7) | Baseline and 3 months
  Changes in overall anxiety will done using the Generalized Anxiety Disorder Questionnaire-7 (GAD-7). The GAD-7 consists of 7 items (scored 0-21) to assess anxiety symptoms over the previous 2 weeks. Higher scores indicate higher frequency of symptoms. Scores greater than or equal to 10 are indicative of generalized anxiety disorder.
Change in overall depression as assessed by the Patient Health Questionnaire-8 (PHQ-8) | Baseline and 3 months
  Changes in overall depression will be assessed using the Patient Health Questionaire-8 (PHQ-8). This consists of a 2-item screen (scored 0-6) from PHQ-2, with a score above 2 prompting PHQ-8. The PHQ-8 consists of 8 items (scored 0-24) to assess depressive symptoms over the previous 2 weeks. Higher scores indicate higher frequency of symptoms, and a score greater than or equal to 10 is indicative of major depression.
Compliance as assessed by the number of patients who consistently used the olfactory training device or solved the Sudoku puzzles | 3 months post intervention
  Patient compliance will be tracked for both groups over the three-month period. Sudoku users will log the number of puzzles completed daily and the time spent on each, while ScentCare users will rely on the companion app to monitor the frequency of their smell training sessions. Compliance data from both methods will be compared after the trial.
Device usability as assessed by the System Usability Scale (SUS) | 3 months post intervention
  Device usability will be evaluated using the System Usability Scale (SUS), a validated 10-item questionnaire. Participants will rate each statement on a scale from 1 (strongly disagree) to 5 (strongly agree). Score range 10-50. Usability scores will be calculated based on SUS guidelines to assess ScentCare's usability and identify areas for improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Rowan, M.D., Principal Investigator — Johns Hopkins University, Department of Otolaryngology - Head and Neck Surgery
Locations (1):
- Johns Hopkins Outpatient Center, Department of Otolaryngology - Head and Neck Surgery, Baltimore, Maryland, United States